CLINICAL TRIAL: NCT02429245
Title: Evaluation of the Accuracy of a Single Cutting Guides System for the Installation of a Total Knee Replacement
Brief Title: Single Cutting Guides System for the Installation of a Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-62
Record Dates: First submitted 2015-04-02; First posted 2015-04-29 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Knee osteoarthritis; Knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Retrospective study

SUMMARY:
The knee prosthesis is a validated treatment for end-stage of knee osteoarthritis, and this intervention usually provides a significant improvement in the quality of life of patients. However, a significant percentage of patients (up to 30%) are disappointed with the outcome of the intervention. One hypothesis that could explain these poor results might be the poor positioning of implants. Individual cutting guides are produced after a CT scan response planning carried out according to the CT scan anatomy of each patient, and subsequently adapted to its real anatomy during surgery, thus theoretically better accuracy of the implementation over conventional techniques. It has been shown in the past that the navigation has been the gold standard in measuring the three-dimensional orientation of the implants during surgery, and this system is systematically used in the service for over 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients operated in the service in 2014 to care for end-stage knee osteoarthritis by implantation of a total knee prosthesis.

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated in the service in 2014 to care for end-stage knee osteoarthritis by implantation of a total knee prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Improvement in the quality of life of patients after Knee replacement | every 3 months over a period of one year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, MD, Principal Investigator — University Hospital, Strasbourg, France

REFERENCES:
- [Derived] De Gori M, Adamczewski B, Jenny JY. Value of the cumulative sum test for the assessment of a learning curve: Application to the introduction of patient-specific instrumentation for total knee arthroplasty in an academic department. Knee. 2017 Jun;24(3):615-621. doi: 10.1016/j.knee.2017.03.007. Epub 2017 Apr 7. PMID 28396050